CLINICAL TRIAL: NCT03243448
Title: Using Skin Sympathetic Nerve Activity to Estimate Sympathetic Tone in Human
Brief Title: Skin Sympathetic Nerve Activity and Sympathetic Tone
Status: Enrolling by invitation | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMU-DK106011
Record Dates: First submitted 2017-07-17; First posted 2017-08-09 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Nerve; Disorder, Sympathetic; Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood sample

GROUPS / COHORTS (2):
- The general public: people between 20-85 years old, without sympathetic hyperactivity disease
- Sympathetic hyperactivity diseases: Sympathetic hyperactivity diseases included: hypertension, heart failure atherosclerotic diseases, arrhythmias, cardiomyopathy, pulmonary hypertension, chronic obstructive pulmonary disease, sleep apnea, pulmonary embolism, hepatitis, liver cirrhosis, hepatopulmonary syndrome, hepatorenal syndrome, renal failure, nephritis, irritable bowel syndrome.

SUMMARY:
There are many sympathetic hyperactivity diseases in the investigators' clinical practice. However, the conventional method to measure the sympathetic nerve activity had many limitations such as clinical application, data interpretation and even therapeutic manipulation. Therefore the investigators would like to develop a non-invasive method to record the sympathetic nerve activity in the investigators' study that can help gathering the sympathetic nerve activity easily in the investigators' daily clinical situation. By the determination of sympathetic nerve activity status, the health caregiver can understand the disease more.

ELIGIBILITY:
Inclusion Criteria:

* Sympathetic hyperactivity diseases included: hypertension, heart failure atherosclerotic diseases, arrhythmias, cardiomyopathy, pulmonary hypertension, chronic obstructive pulmonary disease, sleep apnea, pulmonary embolism, hepatitis, liver cirrhosis, hepatopulmonary syndrome, hepatorenal syndrome, renal failure, nephritis, irritable bowel syndrome.
* Healthy Volunteers

Exclusion Criteria:

* Pregnant

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects who are eligible to the inclusion criteria and admitted to the investigators' ward, visited the investigators' outpatient clinic or health checkup center will be enrolled in the investigators' study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Skin Sympathetic Nerve Activity | 12 hours
  The Sympathetic Nerve Activity Recording from the skin of the subjects in the day time.

SECONDARY OUTCOMES:
ventricular arrhythmia | 24 to 72 hours
  The electrocardiogram recording from the telemetry.
Mortality | 1 to 12 months
  The mortality will be accessed by the chart review and telephone access
Morbidity | 1 to 12 months
  The morbidity will be accessed by the chart review and telephone access

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shen MJ, Coffey AC, Straka S, Adams DE, Wagner DB, Kovacs RJ, Clark M, Shen C, Chen LS, Everett TH 4th, Lin SF, Chen PS. Simultaneous recordings of intrinsic cardiac nerve activity and skin sympathetic nerve activity from human patients during the postoperative period. Heart Rhythm. 2017 Nov;14(11):1587-1593. doi: 10.1016/j.hrthm.2017.06.030. Epub 2017 Jun 23. PMID 28648667
- [Result] Everett TH 4th, Doytchinova A, Cha YM, Chen PS. Recording sympathetic nerve activity from the skin. Trends Cardiovasc Med. 2017 Oct;27(7):463-472. doi: 10.1016/j.tcm.2017.05.003. Epub 2017 May 10. PMID 28619579
- [Result] Uradu A, Wan J, Doytchinova A, Wright KC, Lin AYT, Chen LS, Shen C, Lin SF, Everett TH 4th, Chen PS. Skin sympathetic nerve activity precedes the onset and termination of paroxysmal atrial tachycardia and fibrillation. Heart Rhythm. 2017 Jul;14(7):964-971. doi: 10.1016/j.hrthm.2017.03.030. Epub 2017 Mar 24. PMID 28347833
- [Result] Doytchinova A, Hassel JL, Yuan Y, Lin H, Yin D, Adams D, Straka S, Wright K, Smith K, Wagner D, Shen C, Salanova V, Meshberger C, Chen LS, Kincaid JC, Coffey AC, Wu G, Li Y, Kovacs RJ, Everett TH 4th, Victor R, Cha YM, Lin SF, Chen PS. Simultaneous noninvasive recording of skin sympathetic nerve activity and electrocardiogram. Heart Rhythm. 2017 Jan;14(1):25-33. doi: 10.1016/j.hrthm.2016.09.019. Epub 2016 Sep 23. PMID 27670627
- [Derived] Tang CL, Tsai WC, Lee JY, Wang YK, Chen YH, Liu YW, Lin MC, Fang PT, Huang YL, Wu IC. Higher pre-treatment skin sympathetic nerve activity and elevated resting heart rate after chemoradiotherapy predict worse esophageal cancer outcomes. BMC Cancer. 2022 Oct 22;22(1):1086. doi: 10.1186/s12885-022-10180-8. PMID 36271384
- [Derived] Huang TC, Lin SJ, Chen CJ, Jhuo SJ, Chang CW, Lin SC, Chi NY, Chou LF, Tai LH, Liu YH, Lin TH, Liao WS, Kao PH, Cheng MC, Hsu PC, Lee CS, Lin YH, Lee HC, Lu YH, Yen HW, Lin TH, Su HM, Lai WT, Dai CY, Lee CH, Chen PS, Lin SF, Tsai WC. Skin sympathetic nerve activity and ventricular arrhythmias in acute coronary syndrome. Heart Rhythm. 2022 Oct;19(10):1613-1619. doi: 10.1016/j.hrthm.2022.04.031. Epub 2022 May 5. PMID 35525422